CLINICAL TRIAL: NCT00795626
Title: Impact of Systematic Nursing Orientations in the Reduction of Predicted Cardiovascular Risk in Patients With Coronary Artery Disease.
Acronym: NERE-CR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Eneida Rejane Rabelo da Silva, Professor, PhD., Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UFRGS and HCPA 06570
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Coronary Heart Disease
Keywords: nursing education; cardiovascular risk factors; coronary heart disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle counseling (Experimental): Two groups:
  * control - conventional care
  * intervention - systematic education in the reduction of the risk estimate to cardiovascular events
  Interventions: Behavioral: Systematic education in the reduction of the risk estimate to cardiovascular events

INTERVENTIONS:
Behavioral: Systematic education in the reduction of the risk estimate to cardiovascular events — Systematic education during 4 assessment throughout one year

SUMMARY:
Evaluate the impact of systematic nursing orientations in the reduction of predicted cardiovascular risk in patients with coronary artery disease during four nursing visits for a 1-year period and compare to a group of patients submitted to conventional treatment.

DETAILED DESCRIPTION:
Assess 184 (two groups) patients during four nursing visits for a 1-year period and compare to a group of patients submitted to conventional treatment. We will evaluate the impact of systematic nursing orientations in the reduction of predicted cardiovascular risk in patients with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* patients of both sexes;
* aged 18 years or older;
* diagnosed with ACS (unstable angina and acute myocardial infarction with ST segment elevation and without ST segment elevation) with CAD diagnosed by cardiac catheterization or electrocardiogram;
* patients have to agree to participate by signing a consent term

Exclusion Criteria:

* patients with cognitive deficits;
* neurological sequelae;
* who are not able to come for visits, or who do not consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2007-01; Primary Completion 2011-05 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Reduction of Predicted Cardiovascular Risk | one year

SECONDARY OUTCOMES:
Knowledge of the risk factors and the adhesion to pharmacology treatment; Reduction of the modified risk factors in the previous knowledge of patients and their adhesion; | one year

CONTACTS AND LOCATIONS:
Overall Officials: Eneida R Rabelo, RN, ScD, Principal Investigator — Federal University of Rio Grande do Sul Post Grad Prog
Locations (1):
- Eneida Rejane Rabelo, Porto Alegre, Rio Grande do Sul, Brazil